CLINICAL TRIAL: NCT03894267
Title: An Evaluation of the Impact of a Wound Dressing on Pressure Ulcer Incidence, Among at Risk Individuals, Residing in a Long Stay Health Care Setting (A Pilot RCT Feasibility Study)
Brief Title: An Evaluation of the Impact of a Wound Dressing on Pressure Ulcer Incidence.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NM/1002/2018
Record Dates: First submitted 2018-06-20; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2018-06

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized control design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Self-adhesive silicone bordered foam dressing will be secured to the heels and sacrum.
  Daily SEM reading, visual skin assessment. Early Sense placed under study subject's mattress.
  Follow up 20 days
  Interventions: Device: Cutimed Siltec Heel and Sacrum dressing
- Control Arm (No Intervention): Daily SEM reading, visual skin assessment. Early Sense placed under study subject's mattress.
  Follow up for 20 days.

INTERVENTIONS:
Device: Cutimed Siltec Heel and Sacrum dressing — The dressing has been developed to facilitate exudate management in the treatment of wounds. Newly formed tissue enjoys optimal protection under a moist environment. The foam core with super-absorbers ensures reliable absorption in slightly to heavily exuding wounds. This core has an excellent retention capacity, even under compression. Hydrogen bridges bind the water so securely that, even when subject to pressure, the water is not released. Vertical absorption through the polyurethane foam and the hydro- phobic wound contact layer minimizes the risk of macerations in the peri-ulcer skin.
  Arms: Experimental Arm

SUMMARY:
A pressure ulcer (PU) is localized injury to the skin and/or underlying tissue usually over a bony prominence, as a result of pressure, or pressure in combination with shear. PUs are common, affecting up to 40% of participants receiving health care. Furthermore, PUs impact negatively on an individual's health related quality of life, with pain being the most frequently cited complaint. PUs commonly occur in those who cannot reposition themselves to relieve pressure/shear over bony prominences. The ability to reposition is often diminished in the very old, the malnourished and those with acute illness. Pressure ulcers are common devastating wounds, extending from deep in the bone and muscle layers through to the skin, occurring most often in older persons with limited mobility. They contribute to significant morbidity and mortality as they are smelly, highly painful and very prone to infection.

Existing research carried out by the RCSI School of Nursing and Midwifery shows that both high and low movers are at risk of pressure ulcer development.

DETAILED DESCRIPTION:
A pressure ulcer (PU) is localized injury to the skin and/or underlying tissue usually over a bony prominence, as a result of pressure, or pressure in combination with shear. PUs are common, affecting up to 40% of participants receiving health care. Furthermore, PUs impact negatively on an individual's health related quality of life, with pain being the most frequently cited complaint. PUs commonly occur in those who cannot reposition themselves to relieve pressure/shear over bony prominences. The ability to reposition is often diminished in the very old, the malnourished and those with acute illness. Pressure ulcers are common devastating wounds, extending from deep in the bone and muscle layers through to the skin, occurring most often in older persons with limited mobility. They contribute to significant morbidity and mortality as they are smelly, highly painful and very prone to infection.

Existing research carried out by the RCSI School of Nursing and Midwifery shows that both high and low movers are at risk of pressure ulcer development.

The wound dressing used in this study has been developed to facilitate exudate management in the treatment of wounds. Newly formed tissue enjoys optimal protection under a moist environment. The foam core with super-absorbers ensures reliable absorption in slightly to heavily exuding wounds. This core has an excellent retention capacity, even under compression. Hydrogen bridges bind the water so securely that, even when subject to pressure, the water is not released. Vertical absorption through the polyurethane foam and the hydro- phobic wound contact layer minimizes the risk of macerations in the peri-ulcer skin.

This study is interested in pressure ulcer incidence among low and high movers, residing in a long stay health care facility. The dressing will be applied to intact skin over participant's sacrum and heels as these areas are shown to be at highest risk of pressure ulcer development, in the study population. Participants will be followed up for 20 days, during which time the participant's sacrum and heels will be assessed daily with a non invasive SEM scanner, the EPUAP grading tool, and the usual additional pressure ulcer prevention care. To measure if the participant is a low or high mover an EasySense mobility sensor will be placed under the participant's mattress.

The overall aim of the study is to the impact of the dressing on pressure ulcer incidence in the study population. From a health economics perspective, the management of PUs is suggested to consume 4% of health budgets across Europe, annually. In Ireland PUs of stage 3 and 4 are considered to be serious reportable adverse healthcare events and as such impact negatively on participant safety goals. Furthermore, a recent report from the OECD suggests that PUs are among the most burdensome adverse event type in healthcare, secondary to venous thromboembolism. As such, PUs are a significant threat to participant safety, with prevention being substantially cheaper than treatment5. Indeed, in Europe the cost of PU treatment across all levels of care is estimated at 121.44 million to 2.59 billion EUR, whereas prevention is estimated at 195.27 to 291.33 million EUR5.

ELIGIBILITY:
Inclusion Criteria:

Participants will be considered eligible if they fulfil the following criteria:

* male or female subject aged at least 18 years
* willing and able to give written informed consent and to comply with the requirements
* being at risk of PU development as measured by the activity and mobility components of a mobility assessment tool

Exclusion Criteria:

Participants will be ineligible for enrolment if they meet any of the following criteria:

* unable to provide written informed consent
* known hypersensitivity to any of the ingredients
* participant in any clinical trial of an investigational medicinal product (CTIMP or clinical investigation within 30 days prior to screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Pressure Ulcer incidence | 12 months
  The primary objective is to examine the pressure ulcer occurrence in the two participant groups.

SECONDARY OUTCOMES:
PU incidence related to movement. | 12 months
  The rate of PU incidence among those assessed as high movers compared to those assessed as low movers

CONTACTS AND LOCATIONS:
Overall Officials: Zena Moore, PhD, Principal Investigator — RCSI
Locations (1):
- Cherry Orchard Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Data will be available to other researchers when it is published.